CLINICAL TRIAL: NCT03666884
Title: The Comparison of 50 % Concentration Autologous Serum Eye Drops Versus Preservative Free Artificial Eye Drop Plus 0.05 % Cyclosporin Ophthalmic Emulsion in the Treatment of Severe Dry Eye Syndrome: A Randomized Comparative Study
Brief Title: The Comparison of 50% AS Versus PFAT+ 0.05 % COE in Severe Dry Eye Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seref istek (Other)
Collaborators: Usak State Hospital (Other)
Responsible Party: Sponsor-Investigator, Seref istek, Uşak University Training and Research Hospital, Department of Ophthalmology, Eye Clinic, Principal Investigator, Usak State Hospital
Organization: Usak State Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UsakSH
Record Dates: First submitted 2018-02-20; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Dry Eye Syndrome
Keywords: dry eye; autologous serum; cyclosporine ophthalmic emulsion
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Intervention Model Description: The comparison of 50 % concentration autologous serum eye drops versus preservative free artificial eye drop plus 0.05 % cyclosporin ophthalmic emulsion in the treatment of severe dry eye syndrom
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants chose their treatment regime randomly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- dry eye patients 1 (Active Comparator): dry eye patients treated for 1 month and patient symptoms after 1 month
  Interventions: Drug: COE 2*1 (Restasis) + PFAT Refresh Single dose) 8*1; Biological: AS 50% eye drops 8*1
- dry eye patients 2 (Active Comparator): dry eye patients treated for 1 month and patient symptoms after 1 month
  Interventions: Drug: COE 2*1 (Restasis) + PFAT Refresh Single dose) 8*1; Biological: AS 50% eye drops 8*1

INTERVENTIONS:
Drug: COE 2*1 (Restasis) + PFAT Refresh Single dose) 8*1 — clinical improvement in oxford scale, ocular surface disease index, schirmers test, tear break up time, fluorescein staining of eye
  Other Names: Restasis+Refresh Single Dose
Biological: AS 50% eye drops 8*1 — clinical improvement in oxford scale, ocular surface disease index, schirmers test, tear break up time, fluorescein staining of eye
  Other Names: 50% autologous serum eye drops 8*1

SUMMARY:
The present study aimed to evaluate and compare the efficacy of a 1 month clinical trial of 50% AS for the treatment of severe dry eye syndrom (DES) based on Schirmer's Test, tear break-up time (TBUT), fluorescein staining, and ocular surface disease index (OSDI) scores, as compared to conventional preservative-free artificial tears (PFAT) plus 0.05% COE treatment in patients with severe DES

DETAILED DESCRIPTION:
This is an retrospective comparative study. The designation of the patient whether to use AS 8*1 or conventional PFAT 8*1 plus COE 2*1 was determined randomly. Student's paired samples t-test, independent samples Student's t-test, Wilcoxon signed-rank test and Mann-Whitney U test were used to compare data. All patients responded well to both treatments after the first 1-month treatment period, based on comparison of before and after treatment OSDI scores, Schirmer's test results, TBUT values, and OXFORD scale scores.

ELIGIBILITY:
Inclusion Criteria:

* refractory to conventional treatment (those that did not respond well to entire dry eye medications containing hydroxypropyl methylellulose, carboxyl methylcellulose, polyvinyl alcohol, polyethylene glycol-propylene glycol, sodium hyaluronate, mineral oil, dextran, and carbomer artificial tears with or without preservatives)
* had low TBUT (< 5 s) (5μL of fluorescein sodium 2% eye drops was used)
* low Schirmer's test I score without topical anesthesia ( basic+reflex secretion), positive corneal and conjunctival fluorescein staining (≥grade 1 according to the OXFORD Scale) (3) and an OSDI score > 40 OSDI was a reliable and valid test for quantifying the severity of dry eye symptoms

Exclusion Criteria:

* active ocular infection or any other inflammation not associated with dry eye
* a severe associated ocular allergy, eyelid or eyelash abnormality
* current contact lens use, history of refractive surgery
* associated glaucoma
* current use of any type of topical eye drops other than dry eye medications
* any known graft-versus host disease
* known severe anemia (hemoglobin<11 g/dL-1)
* medically uncontrolled significant cerebrovascular and cardiovascular disease
* pregnant and lactating patients

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10-10 (Actual); Primary Completion 2016-03-15 (Actual); Study Completion 2016-10-25 (Actual)

PRIMARY OUTCOMES:
schirmers test 1 result | first month results after two treatment regimes for severe dry eye groupes, 5 minutes tear drop wetness of schirmers paper in milimeters
  clinical improvement in schirmer's test 1 result
ocular surface oxford scale | first month results after two treatment regimes for severe dry eye groupes, dry eye symptom scale graded 1 to 4
  clinical improvement in oxford scale
ocular surface disease index scale (OSDI) | first month results after two treatment regimes for severe dry eye groupes, dry eye symptoms graduation prepared with sample questions concluded in 2 digit numbers from 25 to 100,
  clinical improvement in OSDI
tear break up time | first month results after two treatment regimes for severe dry eye groupes, dry eye quantitave assesment of tear break up time in seconds graded from 0 sec to 10 seconds 10 the best 0 the worst
  clinical improvement in tear break up time
fluorescein staining of eye | first month results after two treatment regimes for severe dry eye groupes, graduation of dry eye clinical examination graded from 1 to 4
  clinical improvement in fluorescein staining of eye

CONTACTS AND LOCATIONS:
Overall Officials: şeref istek, doctor, Principal Investigator — Department of Ophtalmology, Usak State Hospital

IPD SHARING:
Plan to Share IPD: Yes
study data can be shared
Supporting Information: CSR, Analytic Code
Time Frame: study is finished

REFERENCES:
- [Result] Bradley JC, Bradley RH, McCartney DL, Mannis MJ. Serum growth factor analysis in dry eye syndrome. Clin Exp Ophthalmol. 2008 Nov;36(8):717-20. doi: 10.1111/j.1442-9071.2008.01895.x. PMID 19128374
- [Result] Research in dry eye: report of the Research Subcommittee of the International Dry Eye WorkShop (2007). Ocul Surf. 2007 Apr;5(2):179-93. doi: 10.1016/s1542-0124(12)70086-1. PMID 17508121
- [Result] Bron AJ, Evans VE, Smith JA. Grading of corneal and conjunctival staining in the context of other dry eye tests. Cornea. 2003 Oct;22(7):640-50. doi: 10.1097/00003226-200310000-00008. PMID 14508260
- [Result] Pflugfelder SC, Solomon A, Stern ME. The diagnosis and management of dry eye: a twenty-five-year review. Cornea. 2000 Sep;19(5):644-9. doi: 10.1097/00003226-200009000-00009. PMID 11009316
- [Result] Fox RI, Chan R, Michelson JB, Belmont JB, Michelson PE. Beneficial effect of artificial tears made with autologous serum in patients with keratoconjunctivitis sicca. Arthritis Rheum. 1984 Apr;27(4):459-61. doi: 10.1002/art.1780270415. No abstract available. PMID 6712760
- [Result] Tsubota K, Goto E, Fujita H, Ono M, Inoue H, Saito I, Shimmura S. Treatment of dry eye by autologous serum application in Sjogren's syndrome. Br J Ophthalmol. 1999 Apr;83(4):390-5. doi: 10.1136/bjo.83.4.390. PMID 10434857
- [Result] Lopez-Garcia JS, Garcia-Lozano I, Rivas L, Martinez-Garchitorena J. [Use of autologous serum in ophthalmic practice]. Arch Soc Esp Oftalmol. 2007 Jan;82(1):9-20. doi: 10.4321/s0365-66912007000100004. Spanish. PMID 17262232
- [Result] Rybickova I, Vesela V, Fales I, Skalicka P, Jirsova K. Apoptosis of conjunctival epithelial cells before and after the application of autologous serum eye drops in severe dry eye disease. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2016 Jun;160(2):271-5. doi: 10.5507/bp.2016.001. Epub 2016 Feb 29. PMID 26927466
- [Result] Gao J, Schwalb TA, Addeo JV, Ghosn CR, Stern ME. The role of apoptosis in the pathogenesis of canine keratoconjunctivitis sicca: the effect of topical Cyclosporin A therapy. Cornea. 1998 Nov;17(6):654-63. doi: 10.1097/00003226-199811000-00014. PMID 9820947
- [Result] Ridder WH 3rd. Ciclosporin use in dry eye disease patients. Expert Opin Pharmacother. 2008 Dec;9(17):3121-8. doi: 10.1517/14656560802500613. PMID 19006483
- [Result] Yuksel B, Bozdag B, Acar M, Topaloglu E. Evaluation of the effect of topical cyclosporine A with impression cytology in dry eye patients. Eur J Ophthalmol. 2010 Jul-Aug;20(4):675-9. doi: 10.1177/112067211002000405. PMID 20155706
- [Result] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Result] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Result] Kojima T, Ishida R, Dogru M, Goto E, Matsumoto Y, Kaido M, Tsubota K. The effect of autologous serum eyedrops in the treatment of severe dry eye disease: a prospective randomized case-control study. Am J Ophthalmol. 2005 Feb;139(2):242-6. doi: 10.1016/j.ajo.2004.08.040. PMID 15733983
- [Result] Tananuvat N, Daniell M, Sullivan LJ, Yi Q, McKelvie P, McCarty DJ, Taylor HR. Controlled study of the use of autologous serum in dry eye patients. Cornea. 2001 Nov;20(8):802-6. doi: 10.1097/00003226-200111000-00005. PMID 11685055
- [Result] Leite SC, de Castro RS, Alves M, Cunha DA, Correa ME, da Silveira LA, Vigorito AC, de Souza CA, Rocha EM. Risk factors and characteristics of ocular complications, and efficacy of autologous serum tears after haematopoietic progenitor cell transplantation. Bone Marrow Transplant. 2006 Aug;38(3):223-7. doi: 10.1038/sj.bmt.1705426. Epub 2006 Jun 19. PMID 16785864
- [Result] Welder JD, Bakhtiari P, Djalilian AR. Limbitis secondary to autologous serum eye drops in a patient with atopic keratoconjunctivitis. Case Rep Ophthalmol Med. 2011;2011:576521. doi: 10.1155/2011/576521. Epub 2011 Dec 21. PMID 22606467
- [Result] McDonnell PJ, Schanzlin DJ, Rao NA. Immunoglobulin deposition in the cornea after application of autologous serum. Arch Ophthalmol. 1988 Oct;106(10):1423-5. doi: 10.1001/archopht.1988.01060140587028. PMID 3052385
- [Result] Poon AC, Geerling G, Dart JK, Fraenkel GE, Daniels JT. Autologous serum eyedrops for dry eyes and epithelial defects: clinical and in vitro toxicity studies. Br J Ophthalmol. 2001 Oct;85(10):1188-97. doi: 10.1136/bjo.85.10.1188. PMID 11567963
- [Result] Geerling G, Maclennan S, Hartwig D. Autologous serum eye drops for ocular surface disorders. Br J Ophthalmol. 2004 Nov;88(11):1467-74. doi: 10.1136/bjo.2004.044347. PMID 15489495
- [Result] Cho YK, Huang W, Kim GY, Lim BS. Comparison of autologous serum eye drops with different diluents. Curr Eye Res. 2013 Jan;38(1):9-17. doi: 10.3109/02713683.2012.720340. Epub 2012 Aug 28. PMID 22928476
- [Result] Fischer KR, Opitz A, Boeck M, Geerling G. Stability of serum eye drops after storage of 6 months. Cornea. 2012 Nov;31(11):1313-8. doi: 10.1097/ICO.0b013e3182542085. PMID 22955119
- [Result] Jeng BH, Dupps WJ Jr. Autologous serum 50% eyedrops in the treatment of persistent corneal epithelial defects. Cornea. 2009 Dec;28(10):1104-8. doi: 10.1097/ICO.0b013e3181a2a7f6. PMID 19730088
- [Result] Kojima T, Higuchi A, Goto E, Matsumoto Y, Dogru M, Tsubota K. Autologous serum eye drops for the treatment of dry eye diseases. Cornea. 2008 Sep;27 Suppl 1:S25-30. doi: 10.1097/ICO.0b013e31817f3a0e. PMID 18813071
- [Result] Noble BA, Loh RS, MacLennan S, Pesudovs K, Reynolds A, Bridges LR, Burr J, Stewart O, Quereshi S. Comparison of autologous serum eye drops with conventional therapy in a randomised controlled crossover trial for ocular surface disease. Br J Ophthalmol. 2004 May;88(5):647-52. doi: 10.1136/bjo.2003.026211. PMID 15090417
- [Result] Urzua CA, Vasquez DH, Huidobro A, Hernandez H, Alfaro J. Randomized double-blind clinical trial of autologous serum versus artificial tears in dry eye syndrome. Curr Eye Res. 2012 Aug;37(8):684-8. doi: 10.3109/02713683.2012.674609. Epub 2012 Jun 6. PMID 22670856
- [Result] Ding C, Walcott B, Keyser KT. Sympathetic neural control of the mouse lacrimal gland. Invest Ophthalmol Vis Sci. 2003 Apr;44(4):1513-20. doi: 10.1167/iovs.02-0406. PMID 12657587
- [Result] Stevenson W, Chauhan SK, Dana R. Dry eye disease: an immune-mediated ocular surface disorder. Arch Ophthalmol. 2012 Jan;130(1):90-100. doi: 10.1001/archophthalmol.2011.364. PMID 22232476
- [Result] Sall K, Stevenson OD, Mundorf TK, Reis BL. Two multicenter, randomized studies of the efficacy and safety of cyclosporine ophthalmic emulsion in moderate to severe dry eye disease. CsA Phase 3 Study Group. Ophthalmology. 2000 Apr;107(4):631-9. doi: 10.1016/s0161-6420(99)00176-1. PMID 10768324
- [Result] Kunert KS, Tisdale AS, Gipson IK. Goblet cell numbers and epithelial proliferation in the conjunctiva of patients with dry eye syndrome treated with cyclosporine. Arch Ophthalmol. 2002 Mar;120(3):330-7. doi: 10.1001/archopht.120.3.330. PMID 11879137
- [Result] Kim EC, Choi JS, Joo CK. A comparison of vitamin a and cyclosporine a 0.05% eye drops for treatment of dry eye syndrome. Am J Ophthalmol. 2009 Feb;147(2):206-213.e3. doi: 10.1016/j.ajo.2008.08.015. Epub 2008 Oct 9. PMID 18848318
- [Result] Demiryay E, Yaylali V, Cetin EN, Yildirim C. Effects of topical cyclosporine a plus artificial tears versus artificial tears treatment on conjunctival goblet cell density in dysfunctional tear syndrome. Eye Contact Lens. 2011 Sep;37(5):312-5. doi: 10.1097/ICL.0b013e31822563be. PMID 21792057
- [Result] Stonecipher K, Perry HD, Gross RH, Kerney DL. The impact of topical cyclosporine A emulsion 0.05% on the outcomes of patients with keratoconjunctivitis sicca. Curr Med Res Opin. 2005 Jul;21(7):1057-63. doi: 10.1185/030079905X50615. PMID 16004673
- [Result] Barber LD, Pflugfelder SC, Tauber J, Foulks GN. Phase III safety evaluation of cyclosporine 0.1% ophthalmic emulsion administered twice daily to dry eye disease patients for up to 3 years. Ophthalmology. 2005 Oct;112(10):1790-4. doi: 10.1016/j.ophtha.2005.05.013. PMID 16102833
- [Result] Behrens A, Doyle JJ, Stern L, Chuck RS, McDonnell PJ, Azar DT, Dua HS, Hom M, Karpecki PM, Laibson PR, Lemp MA, Meisler DM, Del Castillo JM, O'Brien TP, Pflugfelder SC, Rolando M, Schein OD, Seitz B, Tseng SC, van Setten G, Wilson SE, Yiu SC; Dysfunctional tear syndrome study group. Dysfunctional tear syndrome: a Delphi approach to treatment recommendations. Cornea. 2006 Sep;25(8):900-7. doi: 10.1097/01.ico.0000214802.40313.fa. PMID 17102664
- [Result] Toshida H, Nguyen DH, Beuerman RW, Murakami A. Neurologic evaluation of acute lacrimomimetic effect of cyclosporine in an experimental rabbit dry eye model. Invest Ophthalmol Vis Sci. 2009 Jun;50(6):2736-41. doi: 10.1167/iovs.08-1880. Epub 2009 Feb 14. PMID 19218606
- [Result] Mah F, Milner M, Yiu S, Donnenfeld E, Conway TM, Hollander DA. PERSIST: Physician's Evaluation of Restasis((R)) Satisfaction in Second Trial of topical cyclosporine ophthalmic emulsion 0.05% for dry eye: a retrospective review. Clin Ophthalmol. 2012;6:1971-6. doi: 10.2147/OPTH.S30261. Epub 2012 Nov 28. PMID 23226002

DOCUMENTS (3):
  • Statistical Analysis Plan (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03666884/SAP_000.pdf
  • Study Protocol (2016-05-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03666884/Prot_001.pdf
  • Informed Consent Form (2015-10-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT03666884/ICF_002.pdf